CLINICAL TRIAL: NCT03225677
Title: Multiple Tracer Using Single Muscle Biopsy Technique in Evaluating Protein Synthesis and Break Down in Muscles of Cirrhotic Patients
Brief Title: Novel Tracer Methods to Evaluate Muscle Protein Metabolism in Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Principal Investigator, The Cleveland Clinic
Other Study IDs: 14-1476
Record Dates: First submitted 2017-04-17; First posted 2017-07-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Cirrhosis: Patients with a diagnosis of cirrhosis will have a blood draw and muscle biopsy will be performed.
  Interventions: Procedure: blood draw and muscle biopsy
- controls: control group should have serum ALT and AST within normal range and a blood draw and muscle biopsy will be performed
  Interventions: Procedure: blood draw and muscle biopsy

INTERVENTIONS:
Procedure: blood draw and muscle biopsy — One venous catheter will be used for bolus injection of multiple labeled AA at the beginning .The second venous catheter will inserted in the other arm for 5 ml of arterialized venous blood draw.Following the infusions, a single muscle biopsy will be performed from the vastus lateralis of the thigh using the Bergstromm needle.

SUMMARY:
To determine the rate and mechanisms of skeletal muscle protein synthesis and breakdown in cirrhotic patients by using multiple tracers and single muscle biopsies.

DETAILED DESCRIPTION:
The goal of this study is to identify the molecular regulatory mechanisms that result in loss of skeletal muscle in cirrhotic patients. Current strategies involve prolonged tracer infusion and multiple muscle biopsies. We will use an innovative approach to determine the rates of skeletal muscle protein synthesis and breakdown using multiple tracers administered at short intervals followed by a single muscle biopsy. These studies are likely to provide a conceptual advance in determining the cellular and molecular responses of the skeletal muscle in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of cirrhosis based on liver biopsy and/or clinical, biochemical, and imaging criteria.
* Patients with Child Pugh score from A5- to B7
* Control group: Subject in control group should have serum ALT and AST within normal range.

Exclusion Criteria for both groups (cirrhotic and control) are:

* diabetes
* cancer
* kidney failure
* pregnancy
* recent surgery (bowel resection or Gastric bypass operation)
* Advanced cardiac or pulmonary disease
* patient with thyroid disease & Coagulopathy ( INR >1.4 and platelet count <80,000/ml)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population: Adults with the diagnosis of cirrhosis will be recruited from the hepatology inpatient service, outpatient clinics and liver transplant clinics at the Cleveland Clinic Foundation. The diagnosis of cirrhosis will be based on liver biopsy and/or clinical, biochemical, and imaging criteria. Will include patient with Child Pugh score from A5- to B7
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Fractional Synthesis Rate | 4 hours
  Fractional synthesis rate (FSR)for each patient is measured by the rate of tracer incorporation from the MIF pool to the bound pool.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Dasarathy, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No